CLINICAL TRIAL: NCT06083233
Title: Role of Brain Specific Biomarkers in Hydrocephalus
Status: Completed | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Miroslav Cihlo, Principal investigator, University Hospital Hradec Kralove
Other Study IDs: MC00002
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hydrocephalus, Normal Pressure; Biochemical Lesions Head Region; Brain Damage
Keywords: Hydrocephalus; Brain biomarkers; Neurofilament Light Chain; Neurofilament Heay Chain; Tau protein; beta-amyloid; Neuron specific enolase; Shunt responsivity
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Brain Injuries; Hydrocephalus; Charcot-Marie-Tooth disease, Type 1F; Frontotemporal Dementia; Plaque, Amyloid | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group "Responders": Patients with diagnosed hydrocephalus undergoing surgery (VP shunt placement) in general anesthesia. Before surgery patients undergo lumbar puncture or external lumbar drainage placement to confirmed the diagnosis and responsivity to VP shunt placement.
  Interventions: Diagnostic Test: Lumbar puncture; Diagnostic Test: External lumbar drainage; Procedure: Ventriculo-peritoneal shunt placement; Procedure: Prechamber puncture; Procedure: Blood sampling #1; Procedure: Blood sampling #2; Procedure: Blood sampling #3; Procedure: Blood sampling #4 and #5
- Study group "Non-responders": Patients with diagnosed hydrocephalus. VP shunt non-responsivity confirmed.
  Interventions: Diagnostic Test: Lumbar puncture; Diagnostic Test: External lumbar drainage; Procedure: Blood sampling #1

INTERVENTIONS:
Diagnostic Test: Lumbar puncture — Standardized lumbar puncture in L3/4 or L4/5 in diagnosis of hydrocephalus and cerebrospinal fluid sampling (sample 1 in measurement)
Diagnostic Test: External lumbar drainage — External lumbar drainage placement for assessing responsivity of external derivation of cerebrospinal fluid. It is test of responsivity to ventriculo-peritoneal shunt placement
Procedure: Ventriculo-peritoneal shunt placement — Surgical procedure based on implantation a thin catheter into brain lateral ventricle (placed through a burrhole from Kocher point) and connection to prechamber and valve (placed behind the ear under skin) and similar thin catheter pushed under skin of neck, chest and abdomen (where put intraperitoneally).
  Groups: Study group "Responders"
Procedure: Prechamber puncture — Puncture of prechamber (place behind the ear under the skin) by thin needle and aspiration of 5 mL of cerebrospinal fluid (5 days, 1 month a 2 months after surgery)
  Groups: Study group "Responders"
Procedure: Blood sampling #1 — Blood sampling to get level of biomarkers (NfL, NfH, NSE, S100, Tau, beta-amyloid) from standardized percutaneous vein puncture by thin needle 24 hours prior surgery
Procedure: Blood sampling #2 — Blood sampling to get level of biomarkers (NfL, NfH, NSE, S100, Tau, beta-amyloid) from standardized percutaneous vein puncture by thin needle 24 hours after surgery
  Groups: Study group "Responders"
Procedure: Blood sampling #3 — Blood sampling to get level of biomarkers (NfL, NfH, NSE, S100, Tau, beta-amyloid) from standardized percutaneous vein puncture by thin needle 5 days after surgery
  Groups: Study group "Responders"
Procedure: Blood sampling #4 and #5 — Blood sampling to get level of biomarkers (NfL, NfH, NSE, S100, Tau, beta-amyloid) from standardized percutaneous vein puncture by thin needle 1 and 2 months after surgery (only in interventional group)
  Groups: Study group "Responders"

SUMMARY:
Normal pressure hydrocephalus (NPH) is a neurodegenerative disease of unclear etiology characterized by a clinical trias named after the neurosurgeon Hakim. It includes cognitive impairment (dementia), gait disturbance, and urinary incontinence. These symptoms, which frequently occur in the elderly population, often overlap with the symptoms of "other" neurodegenerative diseases, especially Alzheimer's disease and other (pre)senile dementias. To distinguishing NPH from "other" dementias is crucial in determining whether a patient will benefit from a surgical procedure (ventriculoperitoneal shunt placement) or not. At the same time, the options for assessing the patient's condition's progression and distinguishing between the progression of neurodegeneration in a broader sense or malfunction of the drainage system are very limited. Therefore, the role of a biomarker that could meet these expectations mentioned above is highly desirable.

DETAILED DESCRIPTION:
Currently, several biomarkers of nerve tissue damage are being studied, which could potentially serve as sensitive and specific biomarkers in the future. These include Neurofilament Light Chain (NfL), Neuron-Specific Enolase (NSE), S100 protein, and tau protein.

A) Neurofilament Light Chain (NfL) and Neurofilament Heavy Chain (NfH):

Neurofilaments (Nfs) are cylindrical proteins found exclusively in neuronal cytoplasm. Under normal conditions, only low levels of the Neurofilament Light Chain (NfL) are released from axons. Elevated levels of NfL have been observed in response to axonal damage in the central nervous system (CNS) due to inflammatory, neurodegenerative, traumatic, or vascular causes, especially in older individuals. NfL is the most soluble subunit of neurofilaments, making its measurement more reliable than other subunits.

The concentration of NfL in cerebrospinal fluid is higher in patients with neurological disorders compared to healthy controls. Similar findings have been reported regarding NfL levels in serum. The role of NfL as a biomarker has been established in conditions such as multiple sclerosis (MS), Alzheimer's disease (AD), frontotemporal dementia (FTD), amyotrophic lateral sclerosis (ALS), atypical parkinsonian disorders (APD), and traumatic brain injury (TBI). It has also been studied to a lesser extent in Creutzfeldt-Jakob disease and neurological complications of HIV infection, where it reaches very high concentrations in cerebrospinal fluid, as well as in Huntington's disease (HD) and normotensive hydrocephalus (NPH or iNPH). Therefore, its implementation in clinical practice is gaining wider acceptance. There is a stronger correlation observed between NfL levels and ALS compared to NfH, although the role of NfH has not been as extensively established yet.

B) Protein S100:

S100 protein belongs to a large family of calcium-binding proteins and is a well-established biomarker in many areas of medicine. In particular, S100B protein is a recognized biomarker in neurodegenerative diseases. Several studies have shown a significant elevation in the levels of S100B in cases of hydrocephalus. However, the relationship between S100B levels and clinical course is not sufficiently explored.

C) Neuron-Specific Enolase (NSE) NSE is an isoenzyme in the glycolytic pathway. Increased levels of NSE have been described in patients with brain injury or stroke. Its half-life in serum is approximately 48 hours. Elevated levels of both S100B and NSE after injuries are associated with an unfavorable outcome and a greater extent of brain tissue damage. In a recent study by Mehmedika-Suljić et al., a non-significantly lower level of NSE was found in patients with hydrocephalus compared to healthy controls. There is a limited number of studies focused on the significance of NSE and its clinical relevance in NPH.

D) Tau Protein and Beta-Amyloid:

There is a close overlap between idiopathic normal pressure hydrocephalus (iNPH) and Alzheimer's disease (AD) because both conditions involve abnormal deposition of toxic byproducts of cerebral metabolism in the brain, such as amyloid-beta 1-42 (amyloid-β 1-42) and Tau protein. Evidence from brain tissue studies even suggests that iNPH could be considered a disease model for Alzheimer's disease. It has also been demonstrated that Alzheimer's disease is a strong predictor of non-responsive iNPH. Recent studies even propose that the final step in neurodegeneration is the pathological cerebral aggregation of toxic brain metabolism byproducts caused by disrupted clearance of these waste products, such as the deposition of amyloid-β 1-42 and Tau in Alzheimer's disease and α-synuclein in Parkinson's disease.

Due to the close association between iNPH and other dementias like Alzheimer's disease and Parkinson's disease, biomarker levels of neurodegeneration in cerebrospinal fluid or blood could potentially be used to differentiate between responsive iNPH and shunt non-responsive iNPH. In this regard, biomarkers such as total Tau (T-Tau) and amyloid-β 1-42 have previously been suggested to assist in this differentiation.

In conclusion, NfL, Tau protein, and beta-amyloid appear to be promising biomarkers that, in many cases, fulfill the role of a marker not only for identifying neuronal damage, such as in the case of postoperative delirium, but also for the regular monitoring of their levels. For conditions like multiple sclerosis (MS), regular monitoring of these biomarkers could serve as a guide in treatment monitoring, medication adjustments, or early identification of subclinical disease relapses. This principle could theoretically be applied to other neurodegenerative diseases as well.

According to some authors, these biomarkers seem to be more sensitive and specific for neuronal damage than, for example, C-reactive protein. Therefore, they hold promise not only for treatment monitoring but also as early identifiers of subclinical disease relapse. Available literature does not suggest significant gender variability in these biomarkers. However, there is a known baseline value that varies with age.

Furthermore, all of the mentioned biomarkers have the potential to distinguish between shunt-responsive and non-responsive iNPH, which is a crucial predictive role in the diagnostic and therapeutic process of iNPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed communicating hydrocephalus
* mini-mental state examination test > 10 points
* Absence of any structural lesion on MRI or CT
* Accepted Informed consent

Exclusion Criteria:

* Non-communicating hydrocephalus
* Structural lesion on MRI or CT (tumour, contusion, aneurysm)
* mini-mental state examination test < 10 points
* Life-expectancy shorter than 1 year
* Pre-existing other type of dementia (m. Alzheimer, vascular dementia)
* Surgery lasting more than 120 minutes
* Blood loss more than 500 ml
* Adverse events during general anesthesia: mean arterial pressure < 60 mm Hg more than 5 minutes, arrythmia with need for pharmacological treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspection on normal pressure hydrocephalus based on neurological examination
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of levels of the mentioned biomarkers | 6 month
  Comparison of levels of the mentioned biomarkers between patients with clinically proven shunt-responsive and shunt-nonresponsive hydrocephalus

SECONDARY OUTCOMES:
Comparison of levels of the biomarkers during follow-up | 6 month
  To follow-up the development of the mentioned biomarker levels during follow-up, comparing them to the evolution of the clinical condition, and exploring the correlation between the levels of individual biomarkers in relation to the monitored parameters of the clinical condition (gait measured by 5-meter-walking test, mini-mental state examination, hydrocephalus parameters by computed tomography or magnetic resonance)

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Cihlo, M.D., Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia